CLINICAL TRIAL: NCT04555668
Title: Effect of Global Postural Reeducation Program With Hamstring Stretch for Patients With Low Back Pain
Brief Title: Effect of Global Postural Reeducation (GPR) Program With Hamstring Stretch for Patients With Low Back Pain
Acronym: GPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00238 Maliha Iftikhar
Record Dates: First submitted 2020-09-16; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Back Pain
Keywords: Low Back Pain; Oswestry Disability Index; Numeric Pain Rating Scale; Stretch
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Global Postural Reeducation Program (Experimental): Global Postural Reeducation Program with hamstring stretch
  Interventions: Other: Global Postural Reeducation Program
- Hamstring Stretch Program (Active Comparator): Hamstring Stretch Program and Knee -flexor eccentric training
  Interventions: Other: Hamstring Stretch Program

INTERVENTIONS:
Other: Global Postural Reeducation Program — Global Postural Reeducation Program with hamstring stretch The lying posture with flexion of the legs aimed to stretch the posterior chain (upper trapezius, levator scapulae, sub occipital, erector spinae, gluteus maximus, ischio-tibial, triceps surae, and foot intrinsic muscles). The initial position will lying with the hip flexed and progression consisted of increasing hip flexion, knee extension, and dorsiflexion of the ankle All above exercises will be given and to be held for 15 minutes each. 40 min/session, 3 times/week for 6 weeks
  Arms: Global Postural Reeducation Program
Other: Hamstring Stretch Program — Hamstring Stretch Program 3 times for 30 seconds hold, subjects rested for 15 seconds between stretches. Knee -flexor eccentric training to prevent hamstring muscle strain 10-15 rep 40 min/session, 3 times/week for 6 weeks
  Arms: Hamstring Stretch Program

SUMMARY:
The purpose of this study is to find out the additional effect of global re-education program with hamstring stretching in patients with low back pain.

DETAILED DESCRIPTION:
Low back pain (LBP) is a very common health problem worldwide and a major cause of disability which affecting performance at work and general well-being. LBP is a complicated condition which affects the physiological and psychosocial aspects of the patient. The muscles of the low back provide the strength and mobility for all activities of daily living. The purpose of this study is to find out the additional effect of global re-education program with hamstring stretching in patients with low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Females
* 18-35 years
* Low back pain > 3 month
* no exercise for last 6 months

Exclusion Criteria:

* Any diagnosed pathology (disc herniation, lumbar stenosis, spinal deformity, fracture, spondylolisthesis)
* Any lower limb abnormality
* Congenital deformities
* Central or peripheral neurologic signs
* Systemic illness (tumor and rheumatologic diseases),
* Psychiatric and mental deficits
* Diabetic neuropathy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 78 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 6th week
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools. For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5.
  0% to 20%: minimal disability 81%-100% exaggerating symptoms.
Numeric Pain Rating Scale | 6th week
  A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pai
Goniometry | 6th week
  A goniometer is an instrument which measures the available range of motion at a joint.
  A large Universal Goniometer having 12-inch arms and full-circle plastic body will be used for measuring Assisted Range of Motion (AROM) for hamstring length, it is a useful measurement tool that can be used to do the Active knee extension test. An active knee-extension test has been shown to be a reliable method of assessing hamstring tightness and has good intra-tester reliability [intraclass correlation coefficient (ICC): 0.97-0.98]

CONTACTS AND LOCATIONS:
Overall Officials: Nazish Rafique, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Helping hand institute of rehabilitation sciences, Mānsehra, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cuenca-Martinez F, Cortes-Amador S, Espi-Lopez GV. Effectiveness of classic physical therapy proposals for chronic non-specific low back pain: a literature review. Phys Ther Res. 2018 Mar 20;21(1):16-22. doi: 10.1298/ptr.E9937. eCollection 2018. PMID 30050749
- [Background] da Silva DA, de Carvalho MEIM, de Andrade Mesquita LS. Effects of a protocol with manual therapy and postural techniques for non-specific low back pain. Manual Therapy, Posturology & Rehabilitation Journal. 2019;17:0-.
- [Background] Cohen SP, Argoff CE, Carragee EJ. Management of low back pain. BMJ. 2008 Dec 22;337:a2718. doi: 10.1136/bmj.a2718. No abstract available. PMID 19103627
- [Background] Parreira P, Maher CG, Steffens D, Hancock MJ, Ferreira ML. Risk factors for low back pain and sciatica: an umbrella review. Spine J. 2018 Sep;18(9):1715-1721. doi: 10.1016/j.spinee.2018.05.018. Epub 2018 May 21. PMID 29792997
- [Background] Bento TPF, Genebra CVDS, Maciel NM, Cornelio GP, Simeao SFAP, Vitta A. Low back pain and some associated factors: is there any difference between genders? Braz J Phys Ther. 2020 Jan-Feb;24(1):79-87. doi: 10.1016/j.bjpt.2019.01.012. Epub 2019 Feb 13. PMID 30782429
- [Background] Abu-Naser SS, ALDAHDOOH R. Lower back pain expert system diagnosis and treatment. 2016.
- [Background] Krismer M, van Tulder M; Low Back Pain Group of the Bone and Joint Health Strategies for Europe Project. Strategies for prevention and management of musculoskeletal conditions. Low back pain (non-specific). Best Pract Res Clin Rheumatol. 2007 Feb;21(1):77-91. doi: 10.1016/j.berh.2006.08.004. PMID 17350545
- [Background] Abdullah IB, Al-Mutairi MM, Alghubayan MA, Alamir AA, Bu-Jubarah AY, Almajed N, et al. Literature Review on Prevalence, Risk Factors and, Evaluation of Acute Lower Back Pain. International Journal of Pharmaceutical Research & Allied Sciences. 2020;9(1).
- [Background] Manchikanti L. Epidemiology of low back pain. Pain Physician. 2000 Apr;3(2):167-92. PMID 16906196
- [Background] Brighton SW. The management of acute low back pain in adults: a guide for the primary care physician, Part II. South African Family Practice. 2013;55(1):26-32.
- [Background] Paolucci T, Attanasi C, Cecchini W, Marazzi A, Capobianco SV, Santilli V. Chronic low back pain and postural rehabilitation exercise: a literature review. J Pain Res. 2018 Dec 20;12:95-107. doi: 10.2147/JPR.S171729. eCollection 2019. PMID 30588084
- [Background] van Tulder MW, Malmivaara A, Esmail R, Koes BW. Exercise therapy for low back pain. Cochrane Database Syst Rev. 2000;(2):CD000335. doi: 10.1002/14651858.CD000335. PMID 10796344
- [Background] Bonetti F, Curti S, Mattioli S, Mugnai R, Vanti C, Violante FS, Pillastrini P. Effectiveness of a 'Global Postural Reeducation' program for persistent low back pain: a non-randomized controlled trial. BMC Musculoskelet Disord. 2010 Dec 16;11:285. doi: 10.1186/1471-2474-11-285. PMID 21162726
- [Background] Guastala FAM, Guerini MH, Klein PF, Leite VC, Cappellazzo R, Facci LM. Effect of global postural re-education and isostretching in patients with nonspecific chronic low back pain: a randomized clinical trial. Fisioterapia em Movimento. 2016;29(3):515-25.
- [Background] Mistry GS, Vyas NJ, Sheth MS. Comparison of hamstrings flexibility in subjects with chronic low back pain versus normal individuals. J Clin Exp Res. 2014;2(1):85-8.